CLINICAL TRIAL: NCT04929171
Title: The Impact of Nociplastic Pain Features on the Response to Physical Therapy in Patients With Primary Myofascial Pain: A Pilot Study.
Brief Title: Myofascial Pain and Central Sensitization
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, David Kohns, Assistant Professor, University of Michigan
Other Study IDs: HUM00093722
Record Dates: First submitted 2021-06-10; First posted 2021-06-18 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Myofascial Pain; Physical Therapy
MeSH Terms: interventions — Physical Therapy Modalities

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with myofascial pain having centralized pain features: Adult patients with myofascial pain having centralized pain features who will be undergoing physical therapy
  Interventions: Other: Physical Therapy

INTERVENTIONS:
Other: Physical Therapy — Physical therapy for chronic upper quarter myofascial pain syndrome, as prescribed by the patients' physicians

SUMMARY:
This prospective, observational cohort pilot study compared pain phenotyping and functional measures in 30 participants with non-acute neck and/or shoulder girdle pain consistent with primary myofascial pain at 3-months following a physical therapy referral to study the impact of their baseline degree of pain amplification.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking participants
* Diagnosed by their physician with non-acute (more than two weeks) neck and/or shoulder girdle primary myofascial pain
* Referred to a physical therapy treatment.

Exclusion Criteria:

* In an effort to reduce the potential that another medical condition could lead to a secondary myofascial pain response, extensive comorbid exclusion criterion.
* Use of chronic high-dose opioid medication greater than 100 mg oral morphine equivalents per day.
* Individuals receiving or applying for compensation or disability.
* The inability to provide informed consent.
* Severe physical impairment (e.g., blindness, deafness)
* Co-morbid medical condition limiting function (e.g., malignant cancer)
* Reported illicit drug use
* Severe psychiatric condition that would limit judgment.
* Lack of internet access.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants were drawn from new patients evaluated at a tertiary care spine and musculoskeletal clinic.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-05-02 (Actual); Primary Completion 2019-11-23 (Actual); Study Completion 2019-11-23 (Actual)

PRIMARY OUTCOMES:
Change in Neck Disability Index | Baseline to 3 months
  Function neck scale with a total possible score of 50 indicating worse function compared to a score of 0.

SECONDARY OUTCOMES:
Change in PEG Score | Baseline to 3 months
  Multidimensional measure for initial assessment and follow-up of chronic pain in a primary care setting. The average of 3 domains with an averaged score of 0 to 10; 0 means lower pain interference and 10 means higher pain interference with life.

CONTACTS AND LOCATIONS:
Overall Officials: David J Kohnsd, DO, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kohns DJ, Scott R, Castellanos J, Scribner D, Hodges R, Clauw DJ. The impact of nociplastic pain features on the response to physical therapy in patients with primary myofascial pain. J Back Musculoskelet Rehabil. 2022;35(5):1143-1151. doi: 10.3233/BMR-210244. PMID 35213348